CLINICAL TRIAL: NCT02071082
Title: A Phase 3b Open-label Study of the Efficacy and Safety of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Single-Tablet Regimen in HIV-1/Hepatitis B Co-infected Adults
Brief Title: Efficacy and Safety of E/C/F/TAF (Genvoya®) in HIV-1/Hepatitis B Co-infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-292-1249
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2017-10

CONDITIONS: HIV; HBV
Keywords: HIV; HBV; Coinfection
MeSH Terms: conditions — Coinfection | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV treatment-naive and HBV treatment-naive (Experimental): HIV/HBV coinfected participants who are HIV treatment-naive and HBV treatment-naive will receive E/C/F/TAF for 48 weeks.
  Interventions: Drug: E/C/F/TAF
- HIV-suppressed (Experimental): HIV/HBV coinfected participants who are HIV-suppressed will receive E/C/F/TAF for 48 weeks.
  Interventions: Drug: E/C/F/TAF

INTERVENTIONS:
Drug: E/C/F/TAF — E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily with food
  Other Names: Genvoya®

SUMMARY:
This study will assess the efficacy, safety, and tolerability of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) fixed-dose combination (FDC) in human immunodeficiency virus (HIV)/hepatitis B virus (HBV) coinfected adults.

Participants will be enrolled into two cohorts:

* Cohort 1: HIV/HBV coinfected adults who are HIV treatment-naive and HBV treatment-naive
* Cohort 2: HIV/HBV coinfected adults who are HIV-suppressed

ELIGIBILITY:
Key Inclusion Criteria:

* Both Cohorts 1 and 2:

  * The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
  * HIV/HBV co-infected adult males and non-pregnant and non-lactating females
  * No evidence of hepatocellular carcinoma (HCC) or clinical or imaging evidence of cirrhosis (ascites, variceal bleeding, encephalopathy).

    --- Subjects should have documentation of an abdominal ultrasound in the 12 months prior to screening, or an abdominal ultrasound at screening, demonstrating the absence of cirrhosis and HCC.
  * Acute Hepatitis A virus (HAV) immunoglobulin M (IgM) negative
  * Hepatitis C virus (HCV) Ab negative, or HCV Ab positive with negative HCV RNA
  * Hepatitis D virus (HDV) Ab negative, or HDV Ab positive with negative HDV RNA
  * Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min according to the Cockcroft-Gault formula
  * CD4+ count of > 200 cells/μL
  * Chronic HBV infection as defined by

    * HBsAg positive for ≥ 6 months Or
    * HBsAg positive at screening and either hepatitis B e antigen (HBeAg) or HBV DNA positive ≥ 6 months Or
    * At screening: positive total hepatitis B core antibody (HBcAb) and negative immunoglobulin M antibody to hepatitis B core antigen (HBcIgM) antibody, and

      * HBsAg positive, or
      * HBeAg positive, or
      * HBV DNA positive
* Cohort 1 (HIV and HBV treatment naive) only:

  * No current or prior anti-HIV treatment, including antiretroviral medications received for prevention (PrEP), or post exposure prophylaxis (PEP)
  * No current or prior anti-HBV treatment
  * Plasma HIV-1 RNA level ≥ 500 copies/mL at screening
  * Screening HBV DNA ≥ 3 log10 IU/mL and < 9 log10 IU/mL
* Cohort 2 (HIV suppressed) only:

  * Receiving current antiretroviral regimen for at least 4 consecutive months
  * No current or prior regimen containing 3 active anti-HBV agents (i.e. cannot be on tenofovir alafenamide (TDF)/emtricitabine (FTC)/Entecavir or TDF/lamivudine(3TC)/Entecavir)
  * Maintained plasma HIV-1 RNA < 50 copies/mL for 6 consecutive months prior to and at the time of the screening visit. Unconfirmed virologic evaluation of ≥ 50 copies/mL after previously reaching viral suppression (transient detectable viremia, or "blip") and prior to screening is acceptable
  * Documented positive HIV antibody test
  * Screening HBV DNA < 9 log10 IU/mL

Key Exclusion Criteria:

* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance use
* A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive carcinoma.
* Received solid organ or bone marrow transplant
* Any history of, or current evidence of, clinical hepatic decompensation (e.g., ascites, encephalopathy or variceal hemorrhage).
* Significant bone disease (e.g., osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, osteochondroses), or multiple bone fractures
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Day 1
* Subjects on hemodialysis, other forms of renal replacement therapy, or on treatment for underlying kidney diseases (including prednisolone, and dexamethasone)
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements
* Investigational agents (unless approved by Gilead Sciences). Participation in any other clinical trial without prior approval from the sponsor is prohibited while participating in this trial

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2015-01-23 (Actual); Study Completion 2016-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (24):
- United States (21):
  - Spectrum Medical Group, Phoenix, Arizona
  - AHF Research Center, Beverly Hills, California
  - Peter J. Ruane MD, Inc., Los Angeles, California
  - Anthony Mills MD, Inc, Los Angeles, California
  - Whitman Walker Health, Washington D.C., District of Columbia
  - Barry M. Rodwick MD, Clearwater, Florida
  - Gary J Richmond M.D.,P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - AIDS Health Foundation/WPA, Miami Beach, Florida
  - AIDS Research and Treatment Center of the Treasure Coast, Vero Beach, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - Be Well Medical Center PC, Berkley, Michigan
  - KC Care Clinic, Kansas City, Missouri
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Southwest CARE Center, Santa Fe, New Mexico
  - Central Texas Clinical Research, Austin, Texas
  - St. Hope Foundation, Bellaire, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Therapeutic Concepts, Houston, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - Peter Shalit MD, Seattle, Washington
- Canada (2):
  - University Health Network/Toronto General Hospital, Toronto, Ontario
  - Maple Leaf Research/Maple Leaf Medical Clinic, Toronto, Ontario
- Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America and Japan. The first participant was screened on 25 February 2014. The last study visit occurred on 26 October 2016.
Pre-assignment Details: 113 participants were screened.
Groups:
- HIV/HBV Treatment-Naive (Cohort 1): HIV/HBV coinfected participants who were HIV treatment-naive and HBV treatment-naive received elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (Genvoya®; E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablet once daily with food for 48 weeks.
- HIV-Suppressed (Cohort 2): HIV/HBV coinfected participants who were HIV-suppressed received E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food for 48 weeks.
Period: Overall Study
Arm/Group | HIV/HBV Treatment-Naive (Cohort 1) | HIV-Suppressed (Cohort 2)
Started | 4 | 75
Completed | 2 | 68
Not Completed | 2 | 7
Not completed — Enrolled and Never Treated | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrew Consent | 0 | 4
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug.
Groups:
- HIV/HBV Treatment-Naive: HIV/HBV coinfected participants who were HIV treatment-naive and HBV treatment-naive received E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food for 48 weeks.
- HIV-Suppressed: HIV/HBV coinfected participants who were HIV-suppressed received E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed | Total
Number analyzed (Participants) | 3 | 74 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (4.0) | 49 (7.8) | 49 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 6
  Male | 3 | 68 | 71
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 7 | 9
  Black | 0 | 14 | 14
  White | 1 | 50 | 51
  Other | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 12 | 12
  Not Hispanic or Latino | 3 | 62 | 65
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 10 | 10
  United States | 1 | 62 | 63
  Japan | 2 | 2 | 4
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.20 (1.242) | 1.29 (0.068) | 1.41 (0.606)
HIV-1 RNA Category [Number; unit: participants]
  < 50 copies/mL | 0 | 73 | 73
  ≥ 50 copies/mL | 3 | 1 | 4
HBV DNA [Mean (Standard Deviation); unit: log10 IU/mL] | 8.31 (0.416) | 1.49 (0.883) | 1.75 (1.588)
HBV DNA Category [Number; unit: participants]
  < 29 IU/mL | 0 | 64 | 64
  ≥ 29 IU/mL | 3 | 10 | 13
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] | 84 (38.9) | 31 (21.1) | 33 (23.9)
Hepatitis B Surface Antigen Status [Number; unit: participants]
  Positive | 3 | 71 | 74
  Negative | 0 | 3 | 3
Hepatitis B e-Antibody Status [Number; unit: participants]
  Positive | 0 | 26 | 26
  Negative | 3 | 43 | 46
  Borderline | 0 | 5 | 5
Fibrotest® Score [Median (Inter-Quartile Range); unit: units on a scale] — The FibroTest® score is used to assess liver fibrosis. Scores range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis.
  units on a scale | 0.27 [0.16 to 0.28] | 0.35 [0.21 to 0.54] | 0.34 [0.21 to 0.53]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 RNA Level < 50 Copies/mL
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Full Analysis Set: participants who were enrolled, received at least 1 dose of study drug, had at least 1 post-Day 1 plasma HBV DNA or HIV-1 RNA result while on study, and had no major protocol violations from the eligibility criteria.
Measure: Number; unit: percentage of participants
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 72
percentage of participants | 100.0 | 94.4

2. Primary Outcome: Percentage of Participants With Plasma HBV DNA Levels < 29 IU/mL
Description: The percentage of participants with HBV DNA < 29 IU/mL at Week 24 was calculated using the missing = failure method.
Time Frame: Week 24
Population: Full Analysis set
Measure: Number; unit: percentage of participants
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 72
percentage of participants | 33.3 | 86.1

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Level < 50 Copies/mL
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 72
percentage of participants | 66.7 | 91.7

4. Secondary Outcome: Percentage of Participants With Plasma HBV DNA Levels < 29 IU/mL
Description: The percentage of participants with HBV DNA < 29 IU/mL at Week 48 was calculated using the missing = failure method.
Time Frame: Week 48
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 72
percentage of participants | 66.7 | 91.7

5. Secondary Outcome: Percentage of Participants With Normalized Alanine Aminotransferase (ALT) at Week 24
Description: ALT normalization was defined as an ALT value that changed from above the normal range at baseline to within the normal range at the given postbaseline visit.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set who had ALT values above the normal range at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 10
percentage of participants | 100.0 | 50.0

6. Secondary Outcome: Percentage of Participants With Normalized ALT at Week 48
Description: as for outcome 5
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set who had ALT values above the normal range at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 10
percentage of participants | 66.7 | 40.0

7. Secondary Outcome: Percentage of Participants With Seroconversion to Hepatitis B Surface Antibody (Anti-HBs) at Week 24
Description: Seroconversion to antibody is defined as (1) antigen loss and (2) positive postbaseline antibody value. Missing = excluded method.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed who had positive antigen and negative antibody at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 70
percentage of participants | 0 | 1.4

8. Secondary Outcome: Percentage of Participants With Seroconversion to Anti-HBs at Week 48
Description: as for outcome 7
Time Frame: Baseline; Week 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 70
percentage of participants | 0 | 1.4

9. Secondary Outcome: Percentage of Participants With Seroconversion to Hepatitis B e Antibody (Anti-HBe) at Week 24
Description: as for outcome 7
Time Frame: Baseline; Week 24
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 30
percentage of participants | 33.3 | 3.3

10. Secondary Outcome: Percentage of Participants With Seroconversion to Anti-HBe at Week 48
Description: as for outcome 7
Time Frame: Baseline; Week 48
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 30
percentage of participants | 33.3 | 0

11. Secondary Outcome: Change From Baseline in FibroTest® Score at Week 24
Description: The FibroTest® score is used to assess liver fibrosis. Scores range from 0.00 to 1.00, with higher scores indicating a greater degree of fibrosis.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 3 | 67
units on a scale | -0.19 [-0.24 to -0.10] | -0.02 [-0.12 to 0.04]

12. Secondary Outcome: Change From Baseline in FibroTest® Score at Week 48
Description: as for outcome 11
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
Number analyzed (Participants) | 2 | 67
units on a scale | -0.15 [-0.21 to -0.08] | -0.07 [-0.12 to 0.02]

ADVERSE EVENTS:
Time Frame: Up to 126 weeks plus 30 days
Description: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug.
Groups:
- HIV/HBV Treatment-Naive: E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily with food for 48 weeks (HIV treatment-naive and HBV treatment-naive)
- HIV-Suppressed: E/C/F/TAF (150/150/200/10 mg) FDC tablet administered orally once daily with food for 48 weeks (HIV-suppressed)
Arm/Group | HIV/HBV Treatment-Naive | HIV-Suppressed
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/3 | 12/74
Other Adverse Events (participants affected / at risk) | 2/3 | 51/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV/HBV Treatment-Naive (N=3) | HIV-Suppressed (N=74)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Meningitis pneumococcal (Infections and infestations) | 0 | 1
Pneumococcal bacteraemia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIV/HBV Treatment-Naive (N=3) | HIV-Suppressed (N=74)
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 7
Vomiting (Gastrointestinal disorders) | 1 | 2
Pyrexia (General disorders) | 0 | 4
Bronchitis (Infections and infestations) | 0 | 6
Chlamydial infection (Infections and infestations) | 0 | 4
Gonorrhoea (Infections and infestations) | 0 | 4
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 4
Nasopharyngitis (Infections and infestations) | 1 | 9
Sinusitis (Infections and infestations) | 0 | 5
Syphilis (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years